CLINICAL TRIAL: NCT07349953
Title: Estimation of Correlation Betweeen Antropometric Characteristics of Children up to 8 Years and Age-based Formulas for Uncuffed Endotracheal Tube in Elective Intubated Children During General Anesthesia
Brief Title: Correlation Between Anthropometric Characteristics and Age-based Formulas for Uncuffed Pediatric Endotracheal Tube
Status: Completed | Type: Observational
Sponsor: Mother and Child Health Institute of Serbia Dr Vukan Cupic (Other)
Responsible Party: Principal Investigator, Ana Mandras, MD, PhD, Mother and Child Health Institute of Serbia Dr Vukan Cupic
Other Study IDs: 8/148
Record Dates: First submitted 2025-12-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endotracheal Tube; Finger
Keywords: Uncuffed endotracheal tube; age-based formula; Circumference of finger

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peditric patients up to 8 years of age requiuring general anesthesia with endotracheal intubation: All patients were scheduled for surgery and elective intubation. Patient's body weight, height, body mass index, and finger circumference were documented. The tube size was selected based on an appropriate formula. After intubation, the circumference of the index, middle, ring, and little fingers of the right and left hands, as well as the child's body mass and height, were measured. The measurement was performed using a flexible meter at the joint of the palm and the root of the finger. Only one anesthesiologist performed the intubation. If the placement of the tube was difficult or there was no audible air leakage around the tube at an inspiratory pressure > 20cmH2O, the selected tube was replaced with a smaller tube by 0.5 mm. If an audible air leak was documented after intubation at an inspiratory pressure of < 10 mmHg, the tube was replaced with a larger tube by 0.5 mm.

SUMMARY:
The goal of this observational study is to investigate the correlation between anthropometric characteristics, such as finger circumferences, body weight, body height, and body mass index, and age-based formulas for uncuffed tube size in pediatric patients up to 8 years of age.

DETAILED DESCRIPTION:
Patients who met inclusion criteria entered the study. All included patients were premedicated with midazolam 0.1mg/kg IV 30 minutes before general anesthesia. Induction: propofol 2,5mg/kg IV, rocuronium 0,6mg/kg IV, fentanyl 3mcg/kg IV; maintenance: sevoflurane 1vol% - 2vol%, fentanyl 3mcg/kg IV as needed. reversion of neuromuscular block was achieved using sugammadex. Trachea was intubated using direct laryngoscopy. Intubation performed one anesthesiologist with more than 10 years of clinical experience in pediatric anesthesia. Initial choice of endotracheal tube (ET) was based on the size of little finger. Proper position of ET was confirmed with chest auscultation, capnography and capnometry. If placing ET was difficult or air leak was not detected using inspiratory pressure > 25cmH2O,ET was replaced with 0,5mm smaller one. If there was air leak using inspiratory pressure < 10 mmHg ET was replaced with 0.5mm bigger one. All children were ventilated using protective strategy. After intubation, measures were made:

1. Finger's circumference was measured with flexible ruler tape (in millimeters). The tape was wrapped around the base of the finger. Circumferences of index finger, middle finger, ring finger and small finger were documented for each hand.
2. Data of body weight, body height and body mass index were taken from patients history.
3. Sizes of used endotracheal tubes were documented.
4. Calculations of ET tube size using age based formulas were made:

for children over 2 years ID (mm) = god/4+4 for children under 2 years of age ODcal (mm) = 0,00223x age(days)+4.88

ELIGIBILITY:
Inclusion Criteria:

* Age up to 8 years of age;
* Children without congenital and acquired anomalies of the trachea;
* Children in whom tracheal intubation is planned as part of the anesthesia plan

Exclusion Criteria:

* Age over 8 years of age;
* The presence of congenital and acquired anomalies of the trachea;
* Children who are already intubated; and failure to obtain informed consent

Ages: 1 Day to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients in this study were admitted to tertiray medical center for scheduled surgery.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was determining the correlation between the size of the selected tube and the circumference of the little finger of the right and left hand | Day 1

SECONDARY OUTCOMES:
determining the correlation between the size of the selected tube and the circumference of the index finger of the right and left hand | Day 1
determining the correlation between the size of the selected tube and the circumference of the middle finger of the right and left hand | Day 1
Determining the correlation between the size of the selected tube and the circumference of the ring finger of the right and left hand | Day 1
determining the correlation between the size of the selected tube and body weight | Day 1
determining the correlation between the size of the selected tube and body height | Day 1
Determining the frequency of post-treatment complications of hoarseness, cough and sore throat | Day 1
determining the frequency of reintubation | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for mother and child health care, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
IPD can be requested by contacting the principal investigator via email: ana_mandras@yahoo.com
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be available after publishing the paper Start date 1.7.2026.
Access Criteria: Access to the IPD will be available for other researchres who are in the ORCID database

REFERENCES:
- [Result] Park S, Shin SW, Kim HJ, Byeon GJ, Yoon JU, Kim EJ, Kim HY. Choice of the correct size of endotracheal tube in pediatric patients. Anesth Pain Med (Seoul). 2022 Oct;17(4):352-360. doi: 10.17085/apm.22215. Epub 2022 Oct 26. PMID 36317427
- [Result] Zhou M, Xu WY, Xu S, Zang QL, Li Q, Tan L, Hu YC, Ma N, Xia JH, Liu K, Ye M, Pu FY, Chen L, Song LJ, Liu Y, Jiang L, Gu L, Zou Z. Prediction of endotracheal tube size in pediatric patients: Development and validation of machine learning models. Front Pediatr. 2022 Oct 20;10:970646. doi: 10.3389/fped.2022.970646. eCollection 2022. PMID 36340734
- [Result] Hanamoto H, Maegawa H, Inoue M, Oyamaguchi A, Kudo C, Niwa H. Age-based prediction of uncuffed tracheal tube size in children to prevent inappropriately large tube selection: a retrospective analysis. BMC Anesthesiol. 2019 Aug 7;19(1):141. doi: 10.1186/s12871-019-0818-3. PMID 31390987